CLINICAL TRIAL: NCT03901261
Title: Cohort Study of Adult Patients With Down Syndrome at Risk of Developing Alzheimer's Disease
Brief Title: Cohort Study of Adult Patients With Down Syndrome at Risk of Developing Alzheimer's Disease (TriAL21)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Jerome Lejeune (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TriAL21
Record Dates: First submitted 2019-02-04; First posted 2019-04-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Down Syndrome; Alzheimer Disease
Keywords: Down Syndrome; Alzheimer Disease; Marker; Neuropsychological; Prodromal; Risk factors
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease | interventions — Spinal Puncture

STUDY DESIGN:
Intervention Model Description: Interventional prospective monocentric, national open study with single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Down syndrome patients (Experimental)
  Interventions: Procedure: Neuro-imaging, Lumbar puncture

INTERVENTIONS:
Procedure: Neuro-imaging, Lumbar puncture — Optional Lumbar Puncture will be performed at inclusion visit Optional Neuro-Imaging (MRI (Magnetic Resonance Imaging) will be performed within 3 months after inclusion visit

SUMMARY:
TriAL21 study is an interventional, open, one arm, prospective, national and single center study.

A total of 200 patients with Down syndrome, aged 35 years and over, without diagnosis of Alzheimer's disease will be enrolled into the study.

Participating centre is Institut Jérôme Lejeune; outpatient's clinic dedicated to treating patients with cognitive deficiencies of genetic origin including patients with Down syndrome.

DETAILED DESCRIPTION:
The aim of the study is to describe and follow a cohort of patients with Down syndrome without diagnosis of Alzheimer's disease at inclusion, in order to identify factors influencing the age of onset of the disease.

The total study duration will be approximately 4 years.

* Inclusion period : 2 years
* Follow-up period per patient : 2 years

Patients will be then followed during 10 years for routine medical follow-up. In case of Alzheimer's disease onset during this period, all data regarding diagnosis of AD will be collected for the study. Data about dementia evolution and mortality in case of AD diagnosis during the study will also be collected during this follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 35 years old and over ;
* Clinical diagnosis of Down syndrome ;
* Patient attending the geriatric outpatient clinic
* Patient without diagnosis of Alzheimer's disease;
* Patient covered by social welfare;
* Patient himself or legal guardian/representative willing and consenting to participate to the study by giving written informed consent;
* Patients must have a parent, or / and other reliable caregiver who agrees to accompany him/her to all visits, provide information about the patient as required by the protocol. The parent or caregiver must be a constant and reliable informant with sufficient contact with the patient to have detailed knowledge of the patient's adaptive functioning in order to be able to complete the assessments accurately.

Exclusion Criteria:

* Patient presenting a contraindication to MRI in particular carrier of metal implants such as pacemakers;
* Patient presenting a serious, severe or unstable pathology (left to the investigator's discretion) whose nature may interfere with the evaluation parameters;
* Patient without Alzheimer's disease diagnosis but with severe dementia;
* Participation in other clinical trials in the last 3 months prior to the study;
* Pregnant woman.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Age of onset of Alzheimer's disease | 2 years
  age (year)
Gender that could influence the age of onset of the disease as determined by medical record review | 2 years
Level of intellectual diasability that could influence the age of onset of the disease as determined by medical record review | 2 years
Family history of Alzheimer's disease that could influence the age of onset of the disease as determined by medical record review | 2 years
Cardio-vascular risk factors that could influence the age of onset of the disease as determined by medical record review | 2 years
Down syndrome comorbidies that could influence the age of onset of the disease as determined by medical record review | 2 years
Genetic's factor other than APP that could influence the age of onset of the disease as determined by medical record review | 2 years
Head trauma that could influence the age of onset of the disease as determined by medical record review | 2 years
Age of menopause that could influence the age of onset of the disease as determined by medical record review | 2 years

SECONDARY OUTCOMES:
Evaluation of neuropsychological evolution using Katz Index of Independence in Activities of Daily Living (Katz ADL) score | 2 years
  Questionnaire about Activities of Daily Living such as bathing, toileting, continence, dressing, transferring and feeding Scoring : Independence: 1 point - Partial dependence 0.5 point - Full dependence: 0 point
Evaluation of neuropsychological evolution using Lawton-Brody Instrumental Activities of Daily Living scale ( IADL) | 2 years
  Questionnaire about strumental Activities of Daily Living such as ability to use telephone, responsibility for taking medication, travels independently on public transportation, ability to handle finances Scoring : 0 or 1
Evaluation of neuropsychological evolution using Dementia Screening Questionnaire for Individuals with Intellectual Disabilities (DSQIID) score | 2 years
  Dementia Screening for Individuals with Intellectual Disabilities Questionnary is a autonomy and psychobeahavioral questionnaire to gather information from carers of people with Down's syndrome about the symptoms of dementia
Evaluation of neuropsychological evolution using Cambridge Examination for Mental Disorders of Older People with Down's Syndrome and Others with Intellectual Disabilities score | 2 years
  Camdex-Ds. Based on an informant interview to aid the diagnosis of dementia in people with DS according to the DSM-IV et ICD criteria for dementia.
Evaluation of neuropsychological evolution using Cambridge Cognition Examination score | 2 years
  It is part of the CAMDEX-DS. Section 2 involves the direct assessment of patient. It contains seven different subscales and has 46 items. it gives a total score of 108. Decline between assessment at Time 1 and assessment at time 2 in association with CAMDEX confirm or evoque the AD diagnosis.
Evaluation of neuropsychological evolution using Cued Recall test score | 2 years
  It is a memory task. It consists in 12 items accompanied by a unique category cue, presented four a time in three trials. It generates two measures respectively for learning phase and delayed recall: a free recall score/12 and a total score/36 (FRS plus items recalled with cue) for the learnig phase. A free recall (FRS/12) and a total score (FRS plus items recalled with cue /12) for the delayed recall. Number of intrusions will be also recorded.
Evaluation of neuropsychological evolution using Cancellation task | 2 years
  Measure of task accuracy (total number of correct responses, range score 0-16) and total time performance (in seconds) were included in the analyses.
Evaluation of neuropsychological evolution using Leiter III assessment score | 2 years
  It is a nonverbal measure of intelligence & cognitive abilities. It includes four subtests whose raw scores are converted to normalised scaled scores (mean [M] = 10, standard deviation [SD] = 3). It gives an IQ standard score (M = 100; SD = 15).
Identification of prodromal Alzheimer's disease markers using brain imaging | 2 years
  Whole brain volumetry calculation, hippocampus volume calculation, white matter lesions volumetry calculation
Identification of prodromal Alzheimer's disease markers using dosage (pg/mL) of biomarkers in cerebrospinal fluid | 2 years
  1-40 beta-amyloid, 1-42 beta-amyloid, tau, phosphorylated tau
Number of adverse event and serious adverse events related to trial procedures | 2 years
  Adverse events graded 3-4-5 according to CTCAE v5.0
Evaluation of survival assessed by vital status | 2 years
  Date and cause of death

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jérôme Lejeune, Paris, France

REFERENCES:
- [Background] Sinai A, Mokrysz C, Bernal J, Bohnen I, Bonell S, Courtenay K, Dodd K, Gazizova D, Hassiotis A, Hillier R, McBrien J, McCarthy J, Mukherji K, Naeem A, Perez-Achiaga N, Rantell K, Sharma V, Thomas D, Walker Z, Whitham S, Strydom A. Predictors of Age of Diagnosis and Survival of Alzheimer's Disease in Down Syndrome. J Alzheimers Dis. 2018;61(2):717-728. doi: 10.3233/JAD-170624. PMID 29226868
- [Background] McCarron M, McCallion P, Reilly E, Dunne P, Carroll R, Mulryan N. A prospective 20-year longitudinal follow-up of dementia in persons with Down syndrome. J Intellect Disabil Res. 2017 Sep;61(9):843-852. doi: 10.1111/jir.12390. Epub 2017 Jun 29. PMID 28664561
- [Background] Mann DM. Alzheimer's disease and Down's syndrome. Histopathology. 1988 Aug;13(2):125-37. doi: 10.1111/j.1365-2559.1988.tb02018.x. PMID 2971602
- [Background] Coppus A, Evenhuis H, Verberne GJ, Visser F, van Gool P, Eikelenboom P, van Duijin C. Dementia and mortality in persons with Down's syndrome. J Intellect Disabil Res. 2006 Oct;50(Pt 10):768-77. doi: 10.1111/j.1365-2788.2006.00842.x. PMID 16961706
- [Background] Lautarescu BA, Holland AJ, Zaman SH. The Early Presentation of Dementia in People with Down Syndrome: a Systematic Review of Longitudinal Studies. Neuropsychol Rev. 2017 Mar;27(1):31-45. doi: 10.1007/s11065-017-9341-9. Epub 2017 Mar 13. PMID 28289920
- [Background] Neale N, Padilla C, Fonseca LM, Holland T, Zaman S. Neuroimaging and other modalities to assess Alzheimer's disease in Down syndrome. Neuroimage Clin. 2017 Nov 6;17:263-271. doi: 10.1016/j.nicl.2017.10.022. eCollection 2018. PMID 29159043
- [Background] Vemuri P, Jack CR Jr. Role of structural MRI in Alzheimer's disease. Alzheimers Res Ther. 2010 Aug 31;2(4):23. doi: 10.1186/alzrt47. PMID 20807454
- [Background] Lleo A, Cavedo E, Parnetti L, Vanderstichele H, Herukka SK, Andreasen N, Ghidoni R, Lewczuk P, Jeromin A, Winblad B, Tsolaki M, Mroczko B, Visser PJ, Santana I, Svenningsson P, Blennow K, Aarsland D, Molinuevo JL, Zetterberg H, Mollenhauer B. Cerebrospinal fluid biomarkers in trials for Alzheimer and Parkinson diseases. Nat Rev Neurol. 2015 Jan;11(1):41-55. doi: 10.1038/nrneurol.2014.232. Epub 2014 Dec 16. PMID 25511894
- [Background] Hulstaert F, Blennow K, Ivanoiu A, Schoonderwaldt HC, Riemenschneider M, De Deyn PP, Bancher C, Cras P, Wiltfang J, Mehta PD, Iqbal K, Pottel H, Vanmechelen E, Vanderstichele H. Improved discrimination of AD patients using beta-amyloid(1-42) and tau levels in CSF. Neurology. 1999 May 12;52(8):1555-62. doi: 10.1212/wnl.52.8.1555. PMID 10331678
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Deb S, Hare M, Prior L, Bhaumik S. Dementia screening questionnaire for individuals with intellectual disabilities. Br J Psychiatry. 2007 May;190:440-4. doi: 10.1192/bjp.bp.106.024984. PMID 17470960
- [Background] Ball SL, Holland AJ, Huppert FA, Treppner P, Watson P, Hon J. The modified CAMDEX informant interview is a valid and reliable tool for use in the diagnosis of dementia in adults with Down's syndrome. J Intellect Disabil Res. 2004 Sep;48(Pt 6):611-20. doi: 10.1111/j.1365-2788.2004.00630.x. PMID 15312062
- [Background] Kim J, Basak JM, Holtzman DM. The role of apolipoprotein E in Alzheimer's disease. Neuron. 2009 Aug 13;63(3):287-303. doi: 10.1016/j.neuron.2009.06.026. PMID 19679070
- [Background] Carmona-Iragui M, Santos T, Videla S, Fernandez S, Benejam B, Videla L, Alcolea D, Blennow K, Blesa R, Lleo A, Fortea J. Feasibility of Lumbar Puncture in the Study of Cerebrospinal Fluid Biomarkers for Alzheimer's Disease in Subjects with Down Syndrome. J Alzheimers Dis. 2017;55(4):1489-1496. doi: 10.3233/JAD-160827. PMID 27858714